CLINICAL TRIAL: NCT00524433
Title: Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety, and Tolerability of Tezosentan in Patients With Acute Heart Failure.
Brief Title: Tezosentan in the Treatment of Acute Heart Failure
Acronym: VERITAS 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-051-307
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Acute Heart Failure; Acute Decompensation of Chronic Heart Failure; New Onset of Heart Failure
Keywords: acute heart failure; acute decompensation of chronic heart failure; new onset of heart failure; tezosentan; Actelion
MeSH Terms: interventions — tezosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): tezosentan
  Interventions: Drug: tezosentan
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tezosentan — tezosentan delivered i.v. at 20 mL/h (5 mg/h) for 30 min followed by 4 mL/h (1 mg/h) for 23.5 to 71.5 h (24 to 72 h in total)
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The randomized patients with acute heart failure will be stratified based on the presence or absence of a Swan-Ganz catheter and assigned to receive either tezosentan 5 mg/h for the first 30 minutes and 1 mg/h thereafter or matching placebo in a 1:1 manner. The duration of the treatment is 24 hours up to 72 hours. The duration of the follow-up period is 30 days after treatment initiation for death, re-hospitalizations and SAEs followed by a follow-up period of 5 months for vital status.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients 18 years of age or older. 2.Male or non-breast-feeding, non-pregnant female (only females who are post menopausal, surgically sterile or practicing a reliable method of contraception).

  3.Acute heart failure (ischemic or non-ischemic). 4.Randomization within 24 hours of hospitalization (including emergency room stay) for acute heart failure.

  5.Dyspnea at rest as assessed by the patient and breathing rate ³ 24/min (measured during 60 seconds).

  6.At least two out of the following four criteria: · elevated BNP or N terminal pro-BNP (more than three times the upper limit of normal for the site) in patients not treated with nesiritide,· clinical evidence of pulmonary congestion/edema (e.g., rales or crackles more than a third above bases),· evidence of pulmonary congestion on chest X-ray, · left ventricular systolic dysfunction (EF < 40% or wall motion index £ 1.2 within 12 months prior to randomization).

  7.Patients in need of i.v. therapy for acute heart failure and who have received at least one dose of i.v. diuretic within 24 hours prior to study drug initiation (last bolus dose must have been more than 2 hours prior to study drug initiation).

  8.Written informed consent.

Exclusion Criteria:

* Criteria only for patients hemodynamically monitored:

  1. Baseline cardiac index > 2.5 l/min/m2 and/or PCWP < 20 mmHg within 6 hours prior to study drug initiation.

     Criteria for all patients:
  2. Patients not receiving i.v. vasodilators (e.g., nitrates, nitroprusside, nesiritide) at baseline: supine systolic blood pressure < 100 mmHg. Patients receiving i.v. vasodilators (e.g., nitrates, nitroprusside, nesiritide) at baseline: supine systolic blood pressure < 120 mmHg.
  3. Cardiogenic shock within the last 48 hours or evidence of volume depletion.
  4. Ongoing myocardial ischaemia, coronary revascularisation procedure (PCI or CABG) during current admission or planned revascularisation.
  5. ST-segment elevation myocardial infarction or administration of thrombolytic therapy.
  6. Baseline creatinine ≥ 2.5 mg/dl (221 mmol/l).
  7. Baseline hemoglobin < 10 g/dl or a hematocrit < 30%.
  8. Hemodialysis, ultrafiltration or peritoneal dialysis within the last 7 days.
  9. Heart failure due to active myocarditis, obstructive hypertrophic cardiomyopathy, congenital heart disease, restrictive cardiomyopathy or constrictive pericarditis. Heart failure caused by valvular disease.
  10. Acute heart failure associated with uncontrolled hemodynamically relevant atrial fibrillation/flutter or ventricular rhythm disturbances.
  11. Acute heart failure secondary to clinical evidence of digoxin toxicity or any other drug-related toxicity.
  12. Significant chronic and/or acute lung disease that might interfere with the ability to interpret the dyspnea assessments or hemodynamic measurements (e.g., severe chronic obstructive pulmonary disease or acute pneumonia).
  13. Mechanical circulatory or ventilatory support. Prior CPAP use is allowed, if discontinued at least 2 hours prior to study drug initiation.
  14. Acute systemic infection/sepsis or other illness with a life expectancy less than 30 days.
  15. Coronary artery bypass graft, or other cardiac surgery, or major non-cardiac surgery within the last 30 days.
  16. Patients who received another investigational drug within 30 days prior to randomization.
  17. Re-randomization in the current study.
  18. Any factors that might interfere with the study conduct or interpretation of the results such as known drug or alcohol dependence.
  19. Concomitant treatment with cyclosporin A or tacrolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2003-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incidence of death or worsening heart failure | within 7 days following study drug initiation

SECONDARY OUTCOMES:
Patient's dyspnea assessment, measured using a visual analog scale | Over first 24 hours

CONTACTS AND LOCATIONS:
Locations (42):
- United States (16):
  - Oracle Research, Huntsville, Alabama
  - USC Medical Center, Los Angeles, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of Miami-Jackson Memorial Hospital, Miami, Florida
  - University Hospital, Augusta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Medical Research Institute, Slidell, Louisiana
  - Baystate Medical Center-Cardiology Section, Springfield, Massachusetts
  - Elmhurst Hospital Center, Elmhurst, New York
  - Columbia Presbyterian Medical Center-Heart Failure Center, New York, New York
  - New York University School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Baylor College of Medicine - Texas Medical Center, Houston, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Alfred Hospital, Monash University, Central and Eastern School, Prahran, Victoria
  - Concord Repatriation Hospital, Concord NSW
  - Queen Elizabeth Hospital, Woodville SA
- Czechia (5):
  - Faculty Hospital St. Anna, Brno
  - Krajska Nemocnice Liberec, Liberec
  - Klinika Kardiologie IKEM, Prague
  - University Hospital Vinohrady (FNKV), Prague
  - Masaryk Hospital, Ústí nad Labem
- Germany (5):
  - Universitatsklinikum der Humboldt-Universitat Berlin, Campus Charite Mitte, Med. Klinik und Poliklinik, Kardiologie, Berlin
  - Universitat Greifswald, Klinik fur Innere Medizin B, Greifswald
  - Asklepios Klinik Langen, Abteilung fur Innere Medizin, Langen
  - Universitatsklinikum Schleswig Holstein, Medizinische Klinik II, Kardiologie, Lübeck
  - Klinik u. Poliklinik F. Inn. Med. II, Univ. Klinik Regensburg, Regensburg
- Hungary (4):
  - Jahn Ferenc, Delpesti Korhaz, Budapest
  - Polyclinic of the Hospitaler Brothers of St. John of God, Budapest
  - University of Debrecen, Debrecen
  - 2nd Department of Medicine & Cardiology Centre, Szeged
- Italy (2):
  - Cattedra di Cardiologia, c/o Spedali Civili, Brescia
  - Istituto Clinico Humanitas, U.O. Cardiologia Clin. E Insuff. Cardiaca, Rozzano (MI)
- Norway (3):
  - Sentralsykehuset i More og Romsdal, Dept. of Cardiology, Ålesund
  - Aker University Hospital, Div. Cardiology, Oslo
  - Central Hospital in Rogaland, Cardiology Division, Stavanger
- United Kingdom (4):
  - University Department of Medicine, City Hospital, Birmingham
  - Cardiology Department, Bridlington & District Hospital, Bridlington
  - University of Glasgow West, Glasgow
  - Dept. of Medicine & Therapeutics, University of Leicester, Leicester

REFERENCES:
- [Derived] Cotter G, Davison BA, Milo O, Bourge RC, Cleland JG, Jondeau G, Krum H, O'Connor CM, Metra M, Parker JD, Torre-Amione G, van Veldhuisen DJ, Kobrin I, Rainisio M, Senger S, Edwards C, McMurray JJ, Teerlink JR; VERITAS Investigators. Predictors and Associations With Outcomes of Length of Hospital Stay in Patients With Acute Heart Failure: Results From VERITAS. J Card Fail. 2016 Oct;22(10):815-22. doi: 10.1016/j.cardfail.2015.12.017. Epub 2015 Dec 22. PMID 26721775
- [Derived] McMurray JJ, Teerlink JR, Cotter G, Bourge RC, Cleland JG, Jondeau G, Krum H, Metra M, O'Connor CM, Parker JD, Torre-Amione G, van Veldhuisen DJ, Lewsey J, Frey A, Rainisio M, Kobrin I; VERITAS Investigators. Effects of tezosentan on symptoms and clinical outcomes in patients with acute heart failure: the VERITAS randomized controlled trials. JAMA. 2007 Nov 7;298(17):2009-19. doi: 10.1001/jama.298.17.2009. PMID 17986694